CLINICAL TRIAL: NCT00304408
Title: Association Between Clinical Response of Clostridium Difficile Colitis to Treatment and Emergence of Anti-C.Difficile Toxin Antibody
Brief Title: Association Between Response to Treatment of C. Diff Colitis and Anti-C.Diff Toxin Antibody
Status: Completed | Type: Observational
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Daniel Musher, MD, VAHouston
Other Study IDs: H-16383
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Clostridium Enterocolitis; Pseudomembranous Colitis; Antibiotic-Associated Colitis
Keywords: Clostridium difficile
MeSH Terms: conditions — Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is three fold: 1)To collect serum from patients with documented Clostridium difficile infection and test for the presence of antibody to C. difficile toxin at the start and at the end of therapy, and again if a relapse or recurrence occurs. 2)To collect stool samples for test of C. difficile toxin at similar time intervals. 3)To assay random serum samples from the VA lab in order to determine the rate of antibody to C. difficile toxin in our patient population.

DETAILED DESCRIPTION:
Clostridium difficile is the leading cause of nosocomial diarrheal disease associated with antibiotic therapy. This is a debilitating condition with substantial morbidity and mortality that may be around 2-3%. Current recommended therapy for this condition is metronidazole, given orally. Our observations suggest that about 10-20% of patients fail to respond to initial therapy with metronidazole, and 20% relapse after treatment. The reason why some persons are cured whereas others relapse is, at present, unknown. There is a suggestion in the medical literature that recurrent infection is associated with the failure to generate antibody to C. difficile toxin. It is also possible that those patients who become infected lack antibody, whereas others in the population tend to have such antibody. The investigators propose to study our patients at VAMC Houston in order to relate occurrence and/or the failure to respond to therapy or the appearance of recurrent disease to the presence of anti-toxin antibody. The investigators also propose to study sera obtained at random from VAMC patients in order to determine the prevalence of antibody in our patient population.

ELIGIBILITY:
Inclusion Criteria:

* All patients at the Houston VA with documented C. difficile infection

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients positive for C. difficile.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. Debakey VA Medical Center, Houston, Texas, United States